CLINICAL TRIAL: NCT04706780
Title: Hemi-diaphragmatic Paresis After Ultrasound-guided Erector Spinae Plane Block in Carotid Endarterectomy
Brief Title: Hemi-diaphragmatic Paresis After Erector Spinae Plane Block
Status: Terminated | Type: Observational
Why Stopped: insufficient number of patients
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 19/27
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-01

CONDITIONS: Regional Anesthesia; Carotid Endarterectomy
Keywords: Regional anesthesia; Erector spinae plane block; Carotid endarterectomy; Ultrasound guidance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ESP block group: Diaphragmatic excursion was measured using M-mode ultrasound during normal breathing, deep breathing and with the sniff manoeuvre.
  Interventions: Other: ESP block

INTERVENTIONS:
Other: ESP block — ESP block performed using ultrasound guidance. Diaphragmatic excursion was measured using M-mode ultrasound during normal breathing, deep breathing and with the sniff manoeuvre.

SUMMARY:
To assess the incidence of hemi-diaphragmatic paresis following ultrasound-guided erector spinae plane (ESP) block

DETAILED DESCRIPTION:
The ultrasound (USG) guided ESP block was first defined in 2016. With the administration of local anesthesia between the transverse process of the vertebra and the erector spinae muscle, it is stated that the effect mechanism of ESP is that spread blocks the ventral and dorsal rami to the paravertebral area. The aim of the study is to assess the incidence of hemi-diaphragmatic paresis following ultrasound-guided erector spinae plane block.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 85 years
* American Society of Anesthesiology (ASA) I-III
* elective carotid endarterectomy

Exclusion Criteria:

* patient's refusal
* under 18 years of age or over 65 years of age
* ASA IV and above
* known allergy to local anaesthetic drugs
* the block cannot be applied due to bleeding disorders or localized skin infection at the injection site
* history of neurological and/or neuromucular disease
* history of severe bronchopulmonary disease
* a moderate to severe decrease in preoperative pulmonary function, or abnormality in preoperative chest radiography data (pleural effusion, pneumothorax, or hemidiaphragm elevation)
* emergency surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: carotid endarterectomy
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
incidence of hemi-diaphragmatic paresis | 30 minutes
  Diaphragmatic excursion was measured using M-mode ultrasound during normal breathing, deep breathing and with the sniff manoeuvre.

SECONDARY OUTCOMES:
opioid consumption | 1 hour
  intraoperative opioid consumption will be recorded
postoperative analgesia consumption | 24 hours
  postoperative analgesia consumption for 24 hours will be recorded
intraoperative local anesthetic consumption | 1 hour
  amount of intraoperative additional local anesthetic consumption will be recorded
Postoperative Numeric Rating Scale (NRS) score | 24 hours
  postoperative pain assessment will be recorded using NRS score (NRS 0=no pain, NRS 10= most severe possible)

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Karaveli, Principal Investigator — Antalya TRH; Ali Sait Kavaklı, Principal Investigator — Antalya TRH
Locations (1):
- Antalya Training and Research Hospital, Department of Anesthesiology and Reanimation, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ueshima H, Hiroshi O. RETRACTED: Erector spinae plane block for carotid endarterectomy. J Clin Anesth. 2018 Aug;48:11. doi: 10.1016/j.jclinane.2018.04.004. Epub 2018 Apr 21. No abstract available. PMID 29684726 (Retraction: PMID 35551828 J Clin Anesth. 2022 Sep;80:110833)
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016